CLINICAL TRIAL: NCT05083260
Title: A Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetics Study in Parkinson's Disease (PD) Participants Treated With Carbidopa/Levodopa and NE3107
Brief Title: NE3107 Activity and Safety in Patients With Parkinson's Disease Using Levodopa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM201
Record Dates: First submitted 2021-09-23; First posted 2021-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: MDS-UPDRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NE3107 (Experimental): orally administered NE3107 20 mg twice daily (BID)
  Interventions: Drug: NE3107
- placebo (Placebo Comparator): orally administered placebo, twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NE3107 — NE3107 is an investigational orally bioavailable, blood-brain barrier permeable anti-inflammatory agent with a new mechanism of action targeting multiple mechanisms of pathology in Parkinson's disease
  Arms: NE3107
Drug: placebo — Hard gelatin capsule containing only common excipients for oral formulations
  Arms: placebo

SUMMARY:
A 28-day phase 2a, double-blind, placebo-controlled (1:1), multi-center study of 20 mg NE3107, twice daily of safety, potential drug-drug interactions, and MDS-UPDRS defined activity in patients with Parkinson's disease . Study will enroll 40 patients that are currently taking immediate release levodopa/ carbidopa (IRLC) and have a practically defined early morning off-state for IRLC. Day one- baseline UPDRS and IRLC PK sampling; day 2- start NE3107 dosing, assess UPDRS during onset and NE3107 PK sampling, rescue meds as needed after 4 hours; day 3 and 14- NE3107 + IRLC UPDRS assessment and PK sampling; day 28- NE3107 + IRLC UPDRS assessments. Optional overnight stays in clinic prior to Day 1-3, 14, and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 30 and no more 80 years of age
2. Diagnosis of PD consistent with UK Brain Bank Criteria or MDS Research Criteria for the Diagnosis of PD, with bradykinesia and a clear motor response to levodopa
3. Stable doses of all PD medications for at least 4 weeks prior to Screening
4. Carbidopa/levodopa dose of at least 300 mg daily, distributed over a minimum of 3 dosing intervals during waking hours
5. Participants must have history of motor fluctuations with reliable early-morning OFF episodes and a history of a good response to levodopa, in the judgement of the investigator
6. If of reproductive potential, willing and able to use a highly effective form of birth control during the study and for 30 days following last dose of study drug. Examples of highly effective forms of birth control are:

   1. Surgical sterility (via vasectomy, hysterectomy, or bilateral tubal ligation) or postmenopausal status in females
   2. Sexual partner who is sterile or of the same sex
   3. Double-barrier method (any combination of physical and chemical methods)
   4. Intrauterine device in females not containing hormones.
7. Able and willing to comply with study drug administration, scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study
8. Investigational Review Board/Ethics Committee-approved consent form signed and date by the participant
9. Assessed as an appropriate and suitable candidate by the Enrollment Authorization Committee (EAC)

Exclusion Criteria:

1. Diagnosis of secondary or atypical parkinsonism
2. Severe or disabling fluctuations or dyskinesias that would, in the opinion of the investigator, interfere with completion of the study
3. Clinically significant cognitive impairment
4. Clinically significant hallucinations or delusions
5. Clinically significant orthostatic hypotension
6. Currently active major depression as determined by BDI-II score of >19
7. Previous surgical procedure for PD (Duopa, DBS, etc.)
8. History of small bowel or gastric surgery
9. History of clinically significant GI abnormality (inflammatory bowel disease, significant motility disorder or emesis of any cause, etc.)
10. Use of long-acting levodopa formulations (Sinemet CR, ER, Rytary, etc.)
11. Routine use of proton pump inhibitors or H2 blockers
12. Routine use of medications that may influence gastric motility (opiates, TCA antidepressants, anticholinergics, etc.)
13. Other clinically significant medical, surgical, psychiatric, or laboratory abnormality that, in the judgment of the investigator, is likely to interfere with study compliance or assessment of safety or efficacy
14. 14) Evidence of significant hepatic impairment according to Child-Pugh criteria, history of cirrhosis, and/or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2.5 times the upper limit of normal (ULN), evidence of ascites, hepatic encephalopathy, bilirubin greater than 2 mg/dL, albumin less than 2.0 g/dL, and INR of 1.5 and greater
15. Significant renal impairment as determined by creatinine clearance (CrCL) less than or equal to 50 mL/min
16. Participant has an ECG or clinical evidence of potentially unstable heart disease, including the following:

    1. QTcF > 470 msec females; > 450 msec males
    2. Complete right or left bundle branch block
    3. Ischemia or myocardial infarct within 1 year prior to the Screening Visit
    4. Clinically significant atrial or ventricular dysrhythmia; the heart must be in predominantly normal sinus rhythm
    5. Second- or third-degree AV block
    6. Heart failure of NYHA classification III or greater
    7. Serious cardiomyopathy or cardiac structural abnormality
    8. Symptomatic coronary artery or ischemic cardiac disease
    9. Any other cardiac condition that the Investigator feels may predispose the participant to ischemia or arrhythmia.
17. Current (or within past 12 months) diagnosis or history of substance abuse, including alcohol (excluding nicotine or caffeine) by Diagnostic and Statistical Manual of Mental Disorders 5 criteria, or positive urine drug screen for tetrahydrocannabinol or any drugs that may affect participant safety or interfere with efficacy assessments
18. Medical or recreational use of marijuana or CBD within 3 months of the Screening Visit
19. Active suicidal ideation within 1 year prior to Screening Visit as determined by a positive response to Question 4 or 5 on the C-SSRS
20. Currently lactating or pregnant, or planning to become pregnant during the study
21. Current participation in another investigational clinical study and/or receipt of any investigational drug within 90 days prior to screening
22. Prior randomization into this study
23. Diabetes requiring insulin treatment
24. Use of potent CYP3A4 inhibitors clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, and verapamil, and potent CYP2C9 and CYP2C19 inhibitors, amiodarone, fluconazole, miconazole, piperine, fluoxetine, fluvoxamine, and ticlopidine.
25. History of breast cancer
26. History of Covid-19 (SARS-CoV-2) infection within 6-weeks prior to screening. Subjects with unresolved symptoms of Covid-19 infection or ongoing cognitive or other deficits attributable to post-Covid-19, that may affect participant safety or interfere with efficacy assessments, based on the Investigator's clinical judgment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline (day 1) in Motor disease society- Unified Parkinson's disease rating scale Part III total score for the patient in the "off-state" (without L-dopa for previous eight hours) | measured on day 1, 2, 3, 14, and 28
  Unified Parkinson's disease rating scale Part III total score is the cumulative score of a 33 question assessment of disease impact on patient's ability to move, with each part scored on a scale of 0-4, with 0 being no effect of disease and 4 being severe disease. a total score of 0 indicates no disease and a total score of 132 indicates the most severe disease
Change from baseline in the length of time during which L-dopa therapy is ineffective in reducing motor symptoms of disease (OFF time) | off time will be measured/recorded every day from day 2 to day 27
  The total sum of time in which a patient self categorizes themselves as in the "off" state determined by diary entries. 0 hours is the minimum/best score, which indicates continuous L-dopa-like activity for the 24 hour period. 24 hours is the worst score and indicates that there was no L-dopa-like benefit at any time during the 24 hour period.
Change from baseline in average Motor disease society- Unified Parkinson's disease rating scale Part III total score measured over the course of 8 hours after taking L-dopa and/or NE3107 | measured on day 1, 2, 3, 14, and 28
  An average score will be calculated from assessments of the Unified Parkinson's disease rating scale Part III total score, which is the cumulative score of a 33 question assessment of disease impact on patient's ability to move, with each question scored on a scale of 0-4, with 0 being no effect of disease and 4 being severe disease. a total score of 0 indicates no disease and a total score of 132 indicates the most severe disease. Scores will be collected several times during the eight hours following L-dopa and/or NE3107 administration.
Motor disease society- Unified Parkinson's disease rating scale Part I total score | measured on day 1, 2, 3, 14, and 28
  the cumulative score of a 13 question assessment of disease impact on patient's cognitive impairment, with each question scored on a scale of 0-4, with 0 being no effect of disease and 4 being severe disease. a total score of 0 indicates no disease and a total score of 42 indicates the most severe disease. This test asks about the impact of disease on cognition, but does not directly measure cognitive capability.
Motor disease society- Unified Parkinson's disease rating scale Part 2 total score | measured on day 1, 2, 3, 14, and 28
  the cumulative score of a 13 question assessment of disease impact on patient's Motor Aspects of Experiences of Daily Living, with each question scored on a scale of 0-4, with 0 being no effect of disease and 4 being a severe effect. a total score of 0 indicates no disease and a total score of 42 indicates the most severe disease.
Change from baseline in the length of time during which L-dopa-like effects are felt by the patient | baseline and day 1, 2, 3, 14, and 28
  The total sum of time in which a patient self categorizes themselves as in the "on" state, with or without dyskinesia determined by diary entries. 0 hours is the minimum/worst score, which indicates no L-dopa-like activity for the 24 hour period. 24 hours is the best score and indicates that there was no L-dopa-like benefit at any time during the 24 hour period.
change from baseline in L-dopa induced dyskinesia measured with the abnormal involuntary movement scale (AIMS) | AIMS will be measured during the 8 hour period of observation on Day 1, 2, 3, 14, and 28
  AIMS is a 12-item clinician-rated scale to assess severity of dyskinesias (orofacial movements and extremity and truncal movements) in patients taking L-dopa. Questions assess the overall severity, incapacitation, and the patient's level of awareness of the movements, and distress associated with them. Questions are scored from 0 (no symptom) to 4 (severe). the minimum total score of 0 indicates no dyskinesia and the maximum total score of 48 indicates severe dyskinesia.
change from baseline in time to onset of L-dopa-like activity | measured on Day 1, 2, 3, 14, and 28
  Length of time from L-dopa administration to beginning of L-dopa activity producing "on-state". Patient self assessment of the time L-dopa-like activity begins after L-dopa administration. A decrease in the time to onset may shorten the time in the off-state and be considered a patient benefit. An increase in time to onset may lengthen time in the off-state and be considered a general worsening of response to treatment.
Change from baseline in Non-Motor Symptom Assessment Scale for Parkinson Disease (NMSS) | Measured on Day 1, 2, 3, 14, and 28
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients at all stages of PD. For each question, scores of severity (0 to 3, with 0 being none and 3 being major source of distress) and frequency (1 to 4, 1= rarely and 4 = very frequent) are recorded and the product of the two calculated. The sum of the products yields the overall score. The minimum total score of 0 indicates no non-motor symptoms and the maximum score of 360 indicates severe disease.
change in area under the levodopa plasma concentration vs. time curve when administered alone compared to being co-administered with NE3107 | Blood samples will be collected on Day 1, 2, 3, and 14
  the plasma concentration vs time curve for L-dopa will be calculated from the L-dopa concentration in plasma samples collected prior to dosing and at 0.5, 1, 2, 3, 4, and 8 hours after L-dopa administration on days on which NE3107 is not administered (Day 1) and three days on which NE3107 is co-administered (Day 2, 3, and 14). Changes in L-dopa area under the curve could be associated with changes in activity against motor symptoms of disease.
Change in the maximum plasma concentration (Cmax) of levodopa when administered alone compared to being co-administered with NE3107. | Blood samples will be collected on Day 1, 2, 3, and 14
  the maximum plasma concentration for L-dopa will be determined in plasma samples collected prior to dosing and at 0.5, 1, 2, 3, 4, and 8 hours after L-dopa administration on days on which NE3107 is not administered (Day 1) and three days on which NE3107 is co-administered (Day 2, 3, and 14). Changes in L-dopa Cmax could be associated with changes in activity against motor symptoms of disease.
The area under the NE3107 plasma concentration vs. time curve when administered alone compared to being co-administered with | Blood samples will be collected on Day 2, 3, and 14
  the plasma concentration vs time curve for NE3107 will be calculated from the NE3107 concentration in plasma samples collected prior to dosing and at 0.5, 1, 2, 3, 4, and 8 hours
Change in the maximum plasma concentration (Cmax) of NE3107 when administered alone compared to being co-administered with L-dopa | Blood samples will be collected on Day 2, 3, and 14
  the maximum plasma concentration for NE3107 will be determined in plasma samples collected prior to dosing and at 0.5, 1, 2, 3, 4, and 8 hours after NE3107 administration

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinson's Disease & Movement Disorders Center Of Boca Raton, Boca Raton, Florida
  - Velocity, Hallandale, Florida
  - Charter Research, Lady Lake, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - First Excellent Research Group, Miami, Florida
  - First Excellent Research, Miami, Florida
  - EZY Medical Research, Miami, Florida
  - Charter Research, Winter Park, Florida
  - Quest Research Institute, Farmington Hills, Michigan
  - New York Neurology Associates, New York, New York
  - Duke University, Durham, North Carolina
  - M3 Wake Research, Raleigh, North Carolina
  - University of Toledo, Toledo, Ohio
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Inland Northwest Research, Spokane, Washington